CLINICAL TRIAL: NCT05016193
Title: Independent Use of Brain Measurement-Based Rehabilitation System by Stroke Survivors: A Randomized Open Label Phase 1 Clinical Trial With Blinded Evaluation
Brief Title: Independent Use of Brain Measurement-Based Rehabilitation System by Stroke Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Axem Neurotechnology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REB20-1200
Record Dates: First submitted 2021-02-08; First posted 2021-08-23 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2021-08

CONDITIONS: Stroke
Keywords: Rehabilitation; Neurofeedback; Functional near-infrared spectroscopy; Neuroergonomics; Motor cortex; Gamification
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): * Participants will attend 3 assessment sessions: one at the beginning of the study, one after about 3 weeks, and one at the end of the study. These sessions will be conducted by a trained physiotherapist.
  * Participants will be asked to wear the Axem Home prototype headband when doing their daily upper-extremity rehabilitation exercises at home.
  * Participants will perform a short motor assessment while wearing the Axem Home prototype headband once per week.
  Interventions: Device: Axem Home Prototype Device; Behavioral: Rehabilitation Exercise Program
- Control Group (Active Comparator): * Participants will attend 3 assessment sessions: one at the beginning of the study, one after about 3 weeks, and one at the end of the study. These sessions will be conducted by a trained physiotherapist.
  * Participants will be asked to keep track of how many minutes of rehabilitation they have completed as per standard care.
  * Participants will perform a short motor assessment while wearing the Axem Home prototype headband once at the beginning of the study and again at the end of the study during the clinical assessment sessions.
  Interventions: Behavioral: Rehabilitation Exercise Program

INTERVENTIONS:
Device: Axem Home Prototype Device — The Axem Home prototype device is a rehabilitation system designed to be used independently by a stroke survivor to facilitate physical rehabilitation exercises in their home environment. The device uses a functional near-infrared spectroscopy (fNIRS) headband that measures the hemodynamic response to rehabilitation exercises and displays this brain activity information to the user.
  Arms: Intervention Group
Behavioral: Rehabilitation Exercise Program — Individual exercise program prescribed by a therapist in the Early Supported Discharge Program.

SUMMARY:
The Axem Home study is a randomized open label trial analyzing the safety and feasibility of coupling the Axem Home prototype device with exercise to improve motor recovery following a stroke.

DETAILED DESCRIPTION:
The Axem Home study is a randomized, open label, phase I clinical trial evaluating the safety and feasibility of coupling feedback to participants on their levels of sensorimotor brain activity (via the Axem Home prototype device) with exercise rehabilitation. 15 participants will be enrolled in each arm of the study. Both groups will participate in an exercise program, but only one group (the intervention group) will receive the Axem Home prototype device.

Study participants will be evaluated at baseline, after 3 weeks, and after 6 weeks (upon the completion of their time in the Early Supported Discharge program). Evaluators will be blinded as to which group participants are in. The study is constructed with randomization to remove selection and allocation biases.

ELIGIBILITY:
Inclusion Criteria:

* Accepted into the Calgary Stroke Program's Early Supported Discharge program for stroke survivors
* Aged 18 or older
* Visual acuity better than 20/50 in both eyes
* Able to give consent
* Clinician reported upper-extremity movement deficit

Exclusion Criteria:

* Score ≥15 on the PHQ-9
* Score <10 on the MoCA or <20 on the CASP
* Inclusion in another interventional trial
* Have open wounds on their scalp

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events Related to the Axem Home Prototype Device (Safety and Tolerability) | Intervention group only: through study completion, an average of 6 weeks
  The ability of participants in the intervention group to complete the study using the Axem Home prototype device without experiencing an adverse event.
Usability Interview | Intervention group only: once per week for an average of 6 weeks and post-intervention (after study completion, an average of week 6)
  A short, semi-structured interview asking participants in the intervention group for qualitative assessments of various aspects of the Axem Home prototype device software and headband, in order to ascertain any potential areas where either might need to be improved.
Usability Questionnaire | Intervention group only: post-intervention (after study completion, an average of week 6)
  A short questionnaire asking participants in the intervention group to rate various aspects of the Axem Home prototype device with respect to its usability and perceived usefulness.
Participation | Intervention group only: through study completion, an average of 6 weeks
  The number of participants in the intervention group that choose to discontinue participation in the study without experiencing an adverse event.

SECONDARY OUTCOMES:
Change in Fugl-Meyer Assessment (FMA) of Motor Recovery | Baseline, week 3, and post-intervention (after study completion, an average of week 6)
  A stroke-specific, performance-based impairment index. The FMA is designed to assess motor functioning, sensation, balance, joint range of motion and joint pain in patients with post-stroke hemiplegia. Sub-scales include: upper extremity (0-36), wrist (0-10), hand (0-14), coordination/speed (0-6) (which can be combined to form a total motor function score out of 66), and sensation (0-4). Higher scores indicate better performance.
Change in Action Research Arm Test (ARAT) score | Baseline, week 3, and post-intervention (after study completion, an average of week 6)
  The ARAT assesses arm function to determine the quality of the arm movement, and the limitation of activity. The ARAT consists of 4 sub-tests; that examines and individual's grip, grasp, pinch and gross motor movement in order to determine upper extremity function. Objects of varying size, shape, and weight must be either grasped, handled or moved in a specific task in order to evaluate function. Low scores mean worse function with the minimum possible score being 0 and the highest possible score being 57 (normal function).
Stroke Impact Scale (SIS) | Baseline, week 3, and post-intervention (after study completion, an average of week 6)
  Stroke-specific, self-report, health status measure. Assesses multiple domains on a 5-point Likert scale. Domains include: strength (4-20), hand function (5-25), activities of daily living/instrumental activities of daily living (10-50), mobility (9-45), communication (7-35), emotion (9-45), memory and thinking (7-35), and participation (8-40). An extra question asks that the patient rate on a scale from 0 - 100 how much they feel that he/she has recovered from his/her stroke. The 4 physical domains (strength, hand function, mobility and activities of daily living) can be summed together to create a single, physical dimension score (28-140) while all other domains should remain separate. Higher scores indicate better function.
National Institutes of Health Stroke Scale (NIHSS) | Baseline
  A 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. Higher scores indicate greater impairment.
Cognitive Assessment for Stroke Patients (CASP) | Baseline
  A questionnaire designed to measure cognitive function in patients regardless of the presence of aphasia, with lower scores indicating greater impairment.
Patient Health Questionnaire (PHQ-9) | Baseline
  A major depressive disorder sub-scale of the full PHQ; used to provisionally grade depressive symptoms in patients. Higher scores indicate the presence of more severe depression.
Montreal Cognitive Assessment (MoCA) | Baseline
  A cognitive screening test used to assess: short term memory, visuospatial abilities, executive functions, attention, concentration, working memory, language, and orientation to time and place. Higher scores indicate better function.
Snellen Eye Chart Assessment of Visual Acuity | Baseline
  Vision will be screened at study entry using a Snellen Eye chart, with acuity ranging from 20/20 (higher acuity) to 20/200 (lower acuity).
Clinician Assessment of Vision | Baseline
  Vision will be screened at study entry by clinician observation to assess visual fields for the presence of visual neglect.
Functional Independence Measure (FIM) | Baseline and post-intervention (after study completion, an average of week 6)
  The FIM rates subjects on 18 items across many functions such as eating, grooming, bathing and dressing on a scale from 1 (total assistance needed) to 7 (complete independence). Lowest possible score is 18 (lowest independence) and the best possible score is 126 (completely independent). The FIM is the standard measure used by rehabilitation facilities in Canada and the United States to evaluate overall function and burden of care.
Modified Rankin Scale (mRS) | Baseline and post-intervention (after study completion, an average of week 6)
  A disability rating scale from 0 (no symptoms at all) to 6 (deceased).
Thumb Localizing Test | Baseline and post-intervention (after study completion, an average of week 6)
  A standardized assessment of proprioception. Scores range from 1 (no difficulty) to 3 (severe difficulty), with lower scores indicating better function.
Strength | Baseline and post-intervention (after study completion, an average of week 6)
  Strength will be assessed using the Medical Research Council scale for muscles in the upper extremity. Scores range from 0 (no movement observed) to 5 (muscle contracts normally against full resistance).
Modified Ashworth Scale (MAS) | Baseline and post-intervention (after study completion, an average of week 6)
  A strength scale used to assess muscle tone during flexion and extension. Scores range from 0 (no increase in tone) to 4 (affected part(s) rigid in flexion or extension), with lower scores indicating better function.
Functional Near-Infrared Spectroscopy (fNIRS) Measures | Intervention group: baseline, once per week for an average of 6 weeks, and post-intervention (after study completion, an average of week 6). Control group: baseline and post-intervention (after study completion, an average of week 6)
  Brain activity feedback from the motor cortex measured during rehabilitation exercises.
Recording of Assigned Home Exercises | Weekly (for an average of 6 weeks)
  Recording of the specific homework exercises assigned by the therapist that the participant completes throughout the week.
Home Exercise Compliance | Weekly (for an average of 6 weeks)
  Proportion of a given participant's weekly assigned home exercise volume (in minutes) they complete.
Video Capture | Intervention group only: rehabilitation sessions (for an average of 6 weeks)
  This data will be used to confirm that the Axem Home prototype device has been correctly placed and securely fitted on the head, which is an assumption of the analysis of functional near-infrared spectroscopy (fNIRS) measures.
Magnetic Resonance Imaging (MRI) | Images taken from within the first week after stroke; collected during the baseline assessment
  Structural images taken from within the first week after stroke (if available). These images will be used to document lesion location and size, and to provide underlying information about functional connections between brain structures.
Computed Tomography Scan Imaging (CT) | Images taken from within the first week after stroke; collected during the baseline assessment
  Structural images taken from within the first week after stroke (if available). These images will be used to document lesion location and size, and to provide underlying information about functional connections between brain structures.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Dukelow, MD PhD FRCPC, Principal Investigator — University of Calgary
Locations (1):
- Calgary Stroke Program Early Supported Discharge, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mihara M, Hattori N, Hatakenaka M, Yagura H, Kawano T, Hino T, Miyai I. Near-infrared spectroscopy-mediated neurofeedback enhances efficacy of motor imagery-based training in poststroke victims: a pilot study. Stroke. 2013 Apr;44(4):1091-8. doi: 10.1161/STROKEAHA.111.674507. Epub 2013 Feb 12. PMID 23404723